CLINICAL TRIAL: NCT00553553
Title: Efficacy Of IV Morphine vs Remifentanil-Intrathecal Morphine Analgesia During Hepatic Resection Surgery
Brief Title: Efficacy of Multimodal Opioid Therapy During Hepatic Resection Surgery
Acronym: RITM-IVM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Dr. N. J. McDonald, St. Vincent's University Hospital, Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: St. Vincent's Hospital Ireland
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Liver Dysfunction; Pain
Keywords: Intrathecal morphine ITM intravenous morphine remifentanil hepatic resection; Adult; ASA I-III (stable); Liver dysfunction requiring primary parenchymal resection
MeSH Terms: conditions — Liver Diseases; Pain | interventions — Morphine; Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): IV morphine group
  Interventions: Drug: Morphine sulphate
- 2 (Experimental): Remifentanil-intrathecal morphine group
  Interventions: Drug: Morphine hydrochloride, remifentanil hydrochloride

INTERVENTIONS:
Drug: Morphine sulphate — Intravenous morphine titrated up to 0.25 milligrams/kilogram prior to end of resection phase or within first 2 hours of surgery
  Arms: 1
Drug: Morphine hydrochloride, remifentanil hydrochloride — Pre-induction intrathecal morphine HCl (< 3 attempts), single shot via 25 G pencil point spinal needle at 10 micrograms/kilogram
  Intra-operative intravenous remifentanil HCl at titratable dose range 0.1-0.25 micrograms/kilogram/minute until start of wound closure
  Arms: 2

SUMMARY:
The patient population requiring hepatic resection can demonstrate an unpredictable risk of exhibiting peri-operative coagulopathy resulting either from the pre-operative hepatic pathophysiology or volume of parenchymal resection. Choice of analgesia can be severely limited.

Currently, the most commonly described use of combined remifentanil infusion and intrathecal morphine has been in fast-track cardiac surgery. To date, there are no published data describing its use in the context of major hepatobiliary where the investigators predict it may provide adequate analgesia with a lower rate of adverse effects over the first 24 hours after surgery.

DETAILED DESCRIPTION:
Choice of analgesia in hepatic resection surgery can be severely limited. This can depend upon on the pre-operative hepatic pathophysiology or the extent of parenchymal resection, both of which will affect peri-operative hepatic function, capacity for drug handling and risk of coagulopathy. Use of IV morphine during hepatic resection can result in high plasma levels post-operatively due to a reduced rate of morphine metabolism, risking a higher rate of morbidity. However, this remains a mainstay of peri-operative analgesia in combination with controversial non-opioid supplementation (paracetamol, non-steroidal anti-inflammatory drugs).

This study compares the efficacy of IV morphine only versus a combination of pre-incisional intrathecal morphine and intra-operative IV remifentanil. Intrathecal morphine provides the mainstay of post-operative analgesia for 12-24 hours and remifentanil provides profound, titratable intra-operative analgesia until the delayed onset of the intrathecal morphine. We hypothesise that this combination might provide desirable intra-operative haemodynamic conditions and eliminate the post-operative additive effects of long-acting, intra-operative IV opioid and intrathecal morphine. Further, if the dose of intrathecal morphine is adequate, this would result in a low rate of post-operative analgesic supplementation and fewer side effects. The titratable dose range of remifentanil is limited to the lower range found to risk post-operative hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* ASA I, II or stable III
* Undergoing primary elective hepatic resection of < 50% predicted parenchymal resection

Exclusion Criteria:

* Previous major upper GI surgery:

  * liver resection or transplant
  * gastrectomy
  * oesophagectomy
  * Whipple's procedure
* Contraindications to dural puncture:

  * coagulopathy
  * uncorrected anti-coagulant therapy
  * spinal deformity
  * neurological disorder
  * psychiatric disorder
* Morphine allergy
* Co-morbidity predisposing to failure of extubation at conclusion of surgery:

  * severe cardiopulmonary pathology scoring ASA III (unstable)
  * IV
  * V
  * sleep apnoea
  * morbid obesity (BMI > 35)
* Failure to proceed with resection, emergency resection or conversion to > 50% parenchymal resection
* Chronic/intractable pain conditions:

  * requiring long-term high dose analgesia
  * implanted analgesic devices
* Predisposition to severe post-operative nausea and vomiting:

  * motion sickness
  * previous PONV
* Anatomical or physiological indication for rapid sequence induction (relative)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-05 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Opioid-related side effects | First 24 hours post-operatively

SECONDARY OUTCOMES:
IV opioid analgesic supplementation | First 24 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Neil J. McDonald, MB BCh, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St. Vincent's University Hospital, Dublin, County Dublin, Ireland